CLINICAL TRIAL: NCT06843122
Title: Evaluation of the Safety and Efficacy of an Advanced Therapy Medicinal Product Containing Live ASCs in the Treatment of Diabetic Foot Syndrome - a Double-blind, Randomized Study.
Brief Title: Evaluation of the Safety and Efficacy of Live ASCs in the Treatment of Diabetic Foot (FOOTCELL)
Acronym: FOOTCELL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FOOTCELL
Record Dates: First submitted 2024-12-30; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: adipose-derived mesenchymal stem cells; chronic wounds; diabetes; foot ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to one of the following arms: Double administration of ADSC/ASC, single administration of ADSC/ASC or Placebo (control) all in addition to SOC treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A - ADSC/ASC cells in fibrin solution - two times administration of ADSC/ASC (Experimental): Application of allogeneic ADSC stem cells in fibrin gel, to cover wound surface with thin cells layer.
  Therapy is based on standard of care procedure for diabetic foot ulcer treatment combined with application of allogeneic ADSC stem cells in fibrin solution onto the wound surface.
  Interventions: Biological: A - Allogenic ADSC cells in fibrin solution - two times administration ADSC/ASC
- B - ADSC/ASC cells in fibrin solution - one administration of ADSC/ASC, one administration placebo (Experimental): Application of allogeneic ADSC stem cells and placebo in fibrin gel, to cover wound surface with thin cells layer.
  Therapy is based on standard of care procedure for diabetic foot ulcer treatment combined with application of allogeneic ADSC stem cells and placebo in fibrin solution onto the wound surface.
  Interventions: Biological: B - Allogenic ADSC cells in fibrin solution - one time administration of ADSC/ASC, one time of placebo
- C - Standard care in diabetic foot ulcer with aplication of fibrin gel to cover wound surface. (Placebo Comparator): Standard of care procedure for diabetic foot ulcer with aplication of fibrin gel to cover wound surface.
  Application of fibrin gel to cover wound surface.
  Interventions: Other: C - Standard care in diabetic foot ulcer with aplication of fibrin gel to cover wound surface.

INTERVENTIONS:
Biological: A - Allogenic ADSC cells in fibrin solution - two times administration ADSC/ASC — ADSC/ASC will be administered twice, at two-week intervals - during V0 and V2 visits The first dose will be administered one week after the randomisation visit. Control visits after administration will be performed every week, up to V6 visit (up to 6 weeks after V0).
  Arms: A - ADSC/ASC cells in fibrin solution - two times administration of ADSC/ASC
Biological: B - Allogenic ADSC cells in fibrin solution - one time administration of ADSC/ASC, one time of placebo — ADSC/ASC will be administered once, at the time of the second application patients will receive a placebo - during V0 and V2 visits The first dose will be administered one week after the randomisation visit. Control visits after administration will be performed weekly, up to V6 visit (up to 6 weeks after V0)
  Arms: B - ADSC/ASC cells in fibrin solution - one administration of ADSC/ASC, one administration placebo
Other: C - Standard care in diabetic foot ulcer with aplication of fibrin gel to cover wound surface. — Placebo will be administered twice, at two-week intervals - during V0 and V2 visits The first dose will be administered one week after the randomisation visit. Control visits after administration will be performed every week, up to V6 visit (up to 6 weeks after V0).
  Arms: C - Standard care in diabetic foot ulcer with aplication of fibrin gel to cover wound surface.

SUMMARY:
The goal of this study is to investigate the safety and efficacy of allogenic mesenchymal stem cells isolated from adipose tissue as the treatment for chronic wounds in diabetic foot syndrome in a double-blinded three armed setup.

DETAILED DESCRIPTION:
Patients will be randomized and assigned to one of three study groups, and will receive according IMP solutions: 1) two doses of cell solution; 2) one dose of cell solution and one dose of placebo solution; 3) two doses of placebo solutions. During the study Patients will attend to weekly visits for routine monitoring and SOC treatment. The IMP solutions will be administered in two weeks intervals, on day 0 and day 14 of the treatment, and the control visits are scheduled on days 7, 21, 28, 35 and 42 - for a total of 7 visits during the active phase of the study. The follow-up visits will be performed 8, 26 and 52 weeks after the last visit in the active phase (day 42).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years at the time of consent,
2. The patient's psychophysical and legal ability to give informed consent to participate in the study,
3. Signing the informed consent document for participation in the study,
4. Ulcer classified as diabetic foot syndrome (DFS) of neuropathic and/or neuroischemic etiology corresponding to grade IA/IIA and IC/IIC according to the University of Texas classification (Appendix E),
5. Duration of the ulcer not less than 6 weeks,
6. Presence of a wound with an area of 1-25 cm² (after wound debridement),
7. Satisfactory blood supply to the wound area:

   * assessed using transcutaneous oxygen pressure measurement, if its value is not less than 30 mmHg,
   * or measurement of systolic blood pressure at the posterior tibial artery and/or dorsalis pedis artery, which is not less than 50 mmHg, to exclude patients who require revascularization therapy,
8. Glycated hemoglobin (HbA1c) < 11%,
9. General health status of the patient, which in the investigator's opinion allows participation in all study procedures,
10. Use of the wound offloading method recommended by the investigator,
11. Use of effective contraception methods to avoid pregnancy (see also Appendix F) and/or based on the following criteria:

    * a woman who is unable to have children (after a hysterectomy or bilateral oophorectomy or post-menopause, defined as a period of at least 12 months since the last menstrual period) is exempt from pregnancy tests,
    * a woman able to have children with a negative pregnancy test result before the administration of the investigational product on the first day and who agrees to periodic pregnancy testing according to the study protocol and to use highly effective contraceptive methods for one month after the end of the active phase of the study (from V6), or two months after the last administration of the investigational drug (from V2).

Exclusion Criteria:

1. Etiology of the ulcer other than diabetic foot syndrome,
2. Presence of an active infection in the wound at the time of inclusion in the study,
3. Wound area <1 cm² or >25 cm²,
4. The patient was enrolled in another clinical trial within the 4 weeks preceding the qualification for this study.
5. Clinically significant limb ischemia:

   * assessed using transcutaneous oxygen pressure measurement, if its value is lower than 30 mmHg
   * or measurement of systolic blood pressure at the posterior tibial artery and/or dorsalis pedis artery, if it is lower than 50 mmHg,
6. Presence of an active phase of Charcot joint,
7. Suspected osteitis and/or osteomyelitis within the study wound,
8. Revascularization procedure on the affected lower limb within 3 months prior to study inclusion or planned revascularization procedure,
9. Chronic kidney disease with GFR < 20 ml/min,
10. Pregnancy and lactation,
11. Allergy to thrombin,
12. Active venous thrombosis,
13. Systemic diseases in the exacerbation stage (acute or decompensated), including heart, kidney, and liver diseases,
14. Active alcohol disease or addiction to psychoactive substances,
15. Allergies to dressing materials used in the study,
16. Oral/intravenous antibiotic therapy at the time of inclusion in the study,
17. Patient undergoing immunosuppressive therapy, including corticosteroid therapy (within 30 days prior to study inclusion),
18. Active cancer or cancer disease in the last 5 years, excluding locally malignant cancers not involving foot tissues,
19. Presence of known clinically active, uncontrolled infections such as hepatitis B, hepatitis C, HIV, and venereal disease (syphilis),
20. Significant features of malnutrition additionally impairing the healing process, regardless of the cause (albumin < 2.5 g/dl and total protein < 5 g/dl),
21. Hemoglobin levels < 9 g/dl,
22. Serum transaminase (alanine and aspartate) activity higher 3x the upper limit of normal (locally).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in wound size (%) at 6 weeks after first study treatment administration compared to baseline with the actual wound size measured by the independent assessor. | 6 weeks after the first administration
  Percentage change in wound size, measured by an independent assessor using a standardized wound area measurement method. The calculation is based on the difference between the baseline wound size and the wound size at 6 weeks, expressed as a percentage of the baseline value.
Type, frequency and severity of adverse events (assessed according CTCAE v5.0); change from baseline of laboratory parameters and selected vital signs of the participants. | 6 weeks after the first administration
  Adverse events will be assessed based on type, frequency, and severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Changes from baseline in laboratory parameters and selected vital signs will be evaluated using standardized clinical measurement methods.

SECONDARY OUTCOMES:
Early efficacy of the allogenic ADSC/ASC defined as percentage of patients with significant clinical success defined as complete wound closure (100% epithelialization), or partial epithelialization of the wound (>50% epithelialization) | 6 weeks after the first administration
  The percentage of patients achieving significant clinical success, defined as either complete wound closure (100% epithelialization) or partial epithelialization of the wound (>50%). Wound epithelialization will be assessed using standardized wound assessment criteria by an independent assessor.
Long-term efficacy of the allogenic ADSC/ASC defined as percentage of patients with significant clinical success defined as complete wound closure (100% epithelialization), or partial epithelialization of the wound (>50% epithelialization) over time. | Through study completion, an average of 1 year
  The percentage of patients achieving significant clinical success, defined as either complete wound closure (100% epithelialization) or partial epithelialization of the wound (>50%), assessed over time. Wound epithelialization will be evaluated using standardized wound assessment criteria by an independent assessor at predefined time points.
The dynamics of wound healing defined as the time required for patients to reach the wound size reduction thresholds: 50% reduction of the wound; maximum reduction of the wound area (%); complete wound healing . | 6 weeks after the first administration and through study completion, an average of 1 year
  The time required for patients to achieve predefined wound size reduction thresholds, including 50% wound size reduction, maximum wound area reduction (percentage), and complete wound healing (100% epithelialization). Wound size will be measured using standardized wound assessment methods by an independent assessor at predefined time points.
Absolute change in the wound-associated pain perception over time assessed by the patient using visual analogue scale. | 6 weeks after the first administration and through study completion, an average of 1 year
  Evaluation of the wound-associated pain, assessed by the patient using visual analogue scale. The minimum value is 0 and means "no pain" and the maximum value is 10 and means "the worst possible pain". The lower value the better outcome.
Additional safety parameters such as wound infection requiring antibiotic treatment expressed as total number of patients, and number of antibiotic therapies per patient. | 6 weeks after the first administration and through study completion, an average of 1 year .
  The total number of patients with wound infections requiring antibiotic treatment and the number of antibiotic therapy courses per patient. Infections will be assessed based on clinical criteria and standard medical guidelines.
Changes in quality of life parameters assessed by the dedicated QoL questionnaire. | 6 weeks after the first administration and through study completion, an average of 1 year
  Evaluation of the patient's quality of life, assessed by the dedicated QoL questionnaire. The QoL questionnaire consists of 10 questions. Each question is scored 1 to 5. The minimum score is 10 and it means "the best possible state of health", and the maximum score is 50, which means ,,the worst possible state of health".

OTHER OUTCOMES:
Evaluation of the additional safety and efficacy parameters such as the percentage of patients requiring lower or upper limb amputation or the percentage of patients experiencing CVD events (CVD death, hospitalization for CVD reason) | through study completion, an average of 1 year
  The percentage of patients requiring lower or upper limb amputation and the percentage of patients experiencing cardiovascular events (CVD death, hospitalization for CVD reasons). Events will be assessed based on clinical diagnosis and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Beata Mrozikiewicz-Rakowska, Assoc.Prof., Principal Investigator — Bielanski Hospital

IPD SHARING:
Plan to Share IPD: Undecided